CLINICAL TRIAL: NCT05176002
Title: The Safety and Efficacy of Camrelizumab in Combination With Radiotherapy for Neoadjuvant Esophageal Squamous Cell Carcinoma.
Brief Title: Camrelizumab in Combination With Radiotherapy for Neoadjuvant Esophageal Carcinoma.
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIRE UNION
Record Dates: First submitted 2021-11-07; First posted 2022-01-04 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2024-12

CONDITIONS: Esophageal Neoplasm; Immunotherapy; Radiotherapy
Keywords: Esophageal Neoplasm; Immunotherapy; radiotherapy; Surgery; Neoadjuvant therapy
MeSH Terms: conditions — Esophageal Neoplasms | interventions — camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant Camrelizumab combined with radiotherapy group (Experimental)
  Interventions: Drug: Camrelizumab

INTERVENTIONS:
Drug: Camrelizumab — Neoadjuvant Camrelizumab combined with radiotherapy

SUMMARY:
This is an exploratory phase II clinical study designed to evaluate the safety and efficacy of Camrelizumab in combination with standard radiotherapy as preoperative neoadjuvant therapy for patients with resectable esophageal squamous cell carcinoma. In the study, all eligible subjects who meet the inclusion criteria will be enrolled after providing full informed consent and signing the informed consent form. All enrolled patients will undergo radical surgery within 4-8 weeks after completion of neoadjuvant Camrelizumab combined with standard radiotherapy.

The safety evaluation indicators include the incidence of adverse events and the number and proportion of subjects who discontinue treatment due to adverse events. The primary efficacy endpoints are the major pathological response rate and the pathological complete response rate. Based on previous studies, the expected response rate is 40% in the experimental group and 20% in the control group. Using a one-sided alpha level of 0.1 and a beta of 0.2, the calculated total sample size for the single-arm design is 25 patients, with 12 enrolled in the first stage. If 2 or fewer responders are observed in the first stage, the study will be terminated early for futility. If more than 2 responders are observed, the trial will proceed to the second stage. Upon completion of the second stage, if the total number of responders exceeds 7, the treatment will be considered effective. The need for postoperative adjuvant treatment and the specific adjuvant regimen will be determined by the investigator. All subjects are required to complete the postoperative follow-up plan as specified in the study protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent prior to the implementation of any trial-related rocedures;
2. Male or female, ≥18 years of age or ≤75 years of age;
3. Patients with a confirmed diagnosis of esophageal squamous cell carcinoma by pathological histology of the primary site biopsy;
4. Patients who are judged to be operable and in need of neoadjuvant therapy by imaging and esophagoscopy ( cT1b-2N+/ cT3-4aN0-3M0), stage II-IVA;
5. The main body of the patient's tumor is located in the mid- and lower thoracic segment of the esophagus as judged by imaging and esophagoscopy (the central location of the tumor is horizontally below the arch of the odd vein, measured endoscopically ≥ 24 cm from the incisors);
6. There is at least one imaging measurable lesion according to the solid tumor efficacy evaluation criteria (RECIST version 1.1);
7. The patient Have not received any prior antitumor therapy, including but not limited to surgery, radiotherapy, chemotherapy, immunotherapy, targeted therapy, etc.;
8. ECOG score 0-1;
9. Adequate organ function, subjects need to meet the following laboratory indices:

   1. Absolute neutrophil count (ANC) ≥ 1.5x109/L in the last 14 days without granulocyte colony-stimulating factor ；
   2. Platelets ≥ 100 x 109/L in the absence of blood transfusion in the last 14 days；
   3. Hemoglobin >9 g/dL without blood transfusion or erythropoietin in the last 14 days;
   4. Total bilirubin ≤1.5 x upper limit of normal (ULN); or total bilirubin >ULN but direct bilirubin ≤ ULN；
   5. Portaline aminotransferase (AST), alanine aminotransferase (ALT) at ≤2.5×ULN;
   6. blood creatinine ≤ 1.5 x ULN and creatinine clearance (calculated using the Cockcroft-Gault formula) ≥ 60 ml/min;
   7. good coagulation function, defined as international normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 times ULN;
   8. normal thyroid function, defined as thyroid stimulating hormone (TSH) within the normal range. If baseline TSH is outside the normal range, subjects with total T3 (or FT3) and FT4 within the normal range may also be enrolled;
   9. Myocardial enzyme profile within the normal range (simple laboratory abnormalities that are not clinically significant, as determined by the investigator, are also allowed).
10. For female subjects of childbearing potential, a negative urine or serum pregnancy test should be performed within 3 days prior to the first dose of study drug (Cycle 1, Day 1). If a negative urine pregnancy test result cannot be confirmed, a blood pregnancy test will be requested. Non-reproductive females are defined as being at least 1 year post-menopausal or having undergone surgical sterilization or hysterectomy;
11. If there is a risk of conception, all subjects (male or female) are required to use contraception with an annual failure rate of less than 1% throughout the treatment period up to 120 days after the final study drug dose.

Exclusion Criteria:

1. patients with an untreated diagnosis of another malignancy within 5 years prior to the first dose (excluding radically treated basal cell carcinoma of the skin, squamous epithelial carcinoma of the skin, and/or radically resected carcinoma in situ)
2. patients at risk for tracheoesophageal fistula or aortoesophageal fistula
3. currently participating in an interventional clinical study treatment or have received another study drug or been treated with an investigational device within 4 weeks prior to the first dose
4. have received prior therapy with: an anti-PD-1, anti-PD-L1 or anti-PD-L2 drug or a drug targeting another stimulatory or co-suppressive T-cell receptor (e.g., CTLA-4, OX-40, CD137).
5. systemic systemic therapy with a proprietary Chinese medicine or immunomodulatory agent (including thymidine, interferon, interleukin, except for local use to control pleural fluid) with an antitumor indication within 2 weeks prior to the first dose.
6. active autoimmune disease requiring systemic therapy (e.g., with disease-relieving drugs, glucocorticoids, or immunosuppressive agents) that occurred within 2 years prior to the first dose. Alternative therapies (e.g., thyroxine, insulin, or physiologic glucocorticoids for adrenal or pituitary insufficiency) are not considered systemic therapy.
7. is receiving systemic glucocorticoid therapy (excluding nasal spray, inhaled or other routes of topical glucocorticoids) or any other form of immunosuppressive therapy within 7 days prior to the first dose of the study.

   Note: Physiological doses of glucocorticoids (≤10 mg/day of prednisone or equivalent) are permitted.
8. known allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation
9. known hypersensitivity to the active ingredient or excipients of the investigational drug Camrelizumab;
10. those with multiple factors affecting oral drug administration (e.g., inability to swallow, post-gastrectomy, chronic diarrhea, and intestinal obstruction)
11. have not recovered sufficiently from toxicity and/or complications from any intervention prior to initiation of therapy (i.e., ≤ grade 1 or at baseline, excluding malaise or alopecia)
12. known history of human immunodeficiency virus (HIV) infection (i.e., positive for HIV 1/2 antibody) and various viral hepatitis infections
13. live vaccination within 30 days prior to the first dose (Cycle 1, Day 1). Note: Injectable inactivated viral vaccine for seasonal influenza within 30 days prior to the first dose is permitted; however, intranasal administration of live attenuated influenza vaccine is not permitted.
14. women who are pregnant or breastfeeding.
15. Presence of any serious or uncontrollable systemic disease, such as

    1. Resting ECG with significant and severely symptomatic uncontrollable abnormalities in rhythm, conduction or morphology, such as complete left bundle branch block, second degree or greater heart block, ventricular arrhythmia or atrial fibrillation.
    2. Unstable angina, congestive heart failure, chronic heart failure of New York Heart Association (NYHA) classification ≥ 2.
    3. myocardial infarction within 6 months prior to randomization
    4. suboptimal blood pressure control (systolic blood pressure > 140 mmHg and diastolic blood pressure > 90 mmHg)
    5. history of non-infectious pneumonia requiring glucocorticoid therapy within 1 year prior to first dose, or current clinically active interstitial lung disease.
    6. active pulmonary tuberculosis.
    7. the presence of an active or uncontrolled infection requiring systemic therapy
    8. presence of clinically active diverticulitis, abdominal abscesses, gastrointestinal obstruction
    9. the presence of liver disease such as cirrhosis, decompensated liver disease, acute or chronic active hepatitis
    10. poorly controlled diabetes mellitus (fasting blood glucose (FBG) > 10 mmol/L)
    11. urine routine suggesting urine protein ≥++ and confirmed 24-hour urine protein quantification >1.0 g
    12. patients with mental disorders and unable to cooperate with treatment
16. have a medical history or evidence of disease that may interfere with the results of the trial, prevent the subject from participating in the study throughout, abnormal treatment or laboratory test values, or other conditions that the investigator considers unsuitable for enrollment The investigator considers that there are other potential risks unsuitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-11-10 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Camrelizumab in Combination With Radiotherapy for Neoadjuvant Esophageal Carcinoma. | 2 week after operation
  Major pathological remission rate
Safety of Camrelizumab in Combination With Radiotherapy for Neoadjuvant Esophageal Carcinoma. | 2 week after operation
  Number and percentage of cases of all adverse events

SECONDARY OUTCOMES:
Efficacy of Camrelizumab in Combination With Radiotherapy for Neoadjuvant | 2 week after operation
  Complete pathology remission rate

CONTACTS AND LOCATIONS:
Overall Officials: Chun Chen, Dortor, Study Chair — Fujian Medical University Affiliated Union Hospital
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided